CLINICAL TRIAL: NCT00599898
Title: Nifedipine Compared to Atosiban for Treating Preterm Labor. A Randomized Controlled Trial.
Brief Title: Nifedipine Compared to Atosiban for Treating Preterm Labor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Raed Salim (Other)
Responsible Party: Sponsor-Investigator, Raed Salim, MD, HaEmek Medical Center, Israel
Organization: HaEmek Medical Center, Israel (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EMC070048CTIL; same as unique protocol ID
Record Dates: First submitted 2008-01-08; First posted 2008-01-24 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Labor, Premature
Keywords: Preterm labor; Atosiban; Nifedipine
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — atosiban; Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Atosiban
- 2 (Experimental)
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Atosiban — Atosiban group will receive an atosiban bolus (6.75 mg) over 1 min then an intravenous infusion of 300mcg/min for 3 h followed by 100mcg/min for another 45h. If contractions continue or recur within 48 hours or the dilatation of the cervix progresses by 1 cm or more within 48 hours, atosiban will be stopped and the women will receive nifedipine as a 2nd line (see arm 2). If the second line fails and gestational age is less than 28 weeks, indomethacin will be administered as a 3rd line.
  Arms: 1
Drug: Nifedipine — Nifedipine group: the initial dose will be 20 mg (one tab) orally every 20 min for 3 doses. If the contractions is inhibited, a maintenance dose of 20 - 40 mg every 6 h up to 48 h will be followed. If contractions continue or recur within 48 hours or the dilatation of the cervix progresses by 1 cm or more within 48 hours, nifedipine will be stopped and the women will receive atosiban as a 2nd line (see arm 2). If the second line fails and gestational age is less than 28 weeks, indomethacin will be administered as a 3rd line.
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the efficacy and the safety of nifedipine compared to atosiban for treating preterm labor.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age between 24 to 34 weeks which had been documented by a definite LMP and sonography up to 20 weeks.
2. All women fulfilled the criteria of preterm labor. The diagnosis of preterm labor required the presence of 4 uterine contractions or more over 30 minutes, each lasting at least 30 seconds, and documented cervical change. The cervical criteria were met when either of the following was present:

   1. Nulliparous women: a single cervical examination demonstrating dilatation of 0 cm to 4 cm and effacement of at least 50%
   2. Multiparous women: a single cervical examination demonstrating dilatation of 1 cm to 4 cm and effacement of at least 50%.
3. Provision of written informed consent

Exclusion Criteria:

1. Chorioamnionitis
2. Preterm rupture of membranes
3. Vaginal bleeding
4. Major fetal malformations
5. Severe hypertensive disorders
6. Intrauterine growth restriction (< 5th percentile).
7. Non-reassuring fetal heart rate
8. Maternal contraindications

   1. Chronic hypertension
   2. Systolic blood pressure < 90 mmHg
   3. Cardiovascular disease
   4. Elevated hepatic enzymes
9. Congenital or acquired uterine malformation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
delaying labor | for more than 48 hours after starting treatment

SECONDARY OUTCOMES:
drugs side effects | within the first 48 hours after treatment
obstetrical (number of days to delivery, gestational age at delivery, mode of delivery) | within 24 hours after delivery
neonatal (Apgar score, sepsis, IVH, NEC, RDS, DEATH) | within 30 days from delivery

CONTACTS AND LOCATIONS:
Overall Officials: Gali Garmi, MD, Principal Investigator — HaEmek Medical Center, Afula, Israel
Locations (1):
- HaEmek Medical Center, Afula, Israel

REFERENCES:
- [Background] King JF, Flenady V, Papatsonis D, Dekker G, Carbonne B. Calcium channel blockers for inhibiting preterm labour; a systematic review of the evidence and a protocol for administration of nifedipine. Aust N Z J Obstet Gynaecol. 2003 Jun;43(3):192-8. doi: 10.1046/j.0004-8666.2003.00074.x. PMID 14712983
- [Background] Papatsonis DN, Van Geijn HP, Ader HJ, Lange FM, Bleker OP, Dekker GA. Nifedipine and ritodrine in the management of preterm labor: a randomized multicenter trial. Obstet Gynecol. 1997 Aug;90(2):230-4. doi: 10.1016/S0029-7844(97)00182-8. PMID 9241299
- [Background] Moutquin JM, Sherman D, Cohen H, Mohide PT, Hochner-Celnikier D, Fejgin M, Liston RM, Dansereau J, Mazor M, Shalev E, Boucher M, Glezerman M, Zimmer EZ, Rabinovici J. Double-blind, randomized, controlled trial of atosiban and ritodrine in the treatment of preterm labor: a multicenter effectiveness and safety study. Am J Obstet Gynecol. 2000 May;182(5):1191-9. doi: 10.1067/mob.2000.104950. PMID 10819857
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046
- [Derived] Salim R, Garmi G, Nachum Z, Zafran N, Baram S, Shalev E. Nifedipine compared with atosiban for treating preterm labor: a randomized controlled trial. Obstet Gynecol. 2012 Dec;120(6):1323-31. doi: 10.1097/aog.0b013e3182755dff. PMID 23168756